CLINICAL TRIAL: NCT00013325
Title: Cardiac Disease and the Electrocardiogram in SCI Patients
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: B2140R
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2001-01

CONDITIONS: Spinal Cord Injury
Keywords: Spinal cord injury, heart disease, electrocardiography
MeSH Terms: conditions — Spinal Cord Injuries; Heart Diseases

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Cardiac Disease

SUMMARY:
The purpose of this three-year study is to determine the prevalence and incidence of the different types of cardiac disease and ECG abnormalities in SCI patients. Study goals are: (i) delineation of the specific types of heart disease that occur in the SCI population as manifested both pre-clinically and clinically and (ii) demonstration of their association with ECG findings. This will enable validation of scores and algorithms using the inexpensive and widely available ECG for the prevention of heart disease as well as it's early treatment and rehabilitation in SCI patients.

The findings will be helpful in demonstrating what cardiological tests are appropriate for the mandated annual evaluation of SCI patients.

DETAILED DESCRIPTION:
The purpose of this three-year study is to determine the prevalence and incidence of the different types of cardiac disease and ECG abnormalities in SCI patients seen at the PAVA SCIC and their association. Study goals include: i) delineation of the specific types of heart disease that occur in the SCI population as manifested both pre-clinically and clinically and ii) demonstration of their association with ECG findings. This will enable validation of scores and algorithms using the inexpensive and widely available ECG for the prevention of heart disease as well as it's early treatment and rehabilitation in SCI patients. Our findings will be helpful in demonstrating what cardiological tests are appropriate for the mandated annual evaluation of SCI patients.

There are two components to this study:

An outcomes component to complete information previously gathered in clinical and computerized databases of 800 SCI patients and a convenience sample of age-matched able-bodied veterans and perform a follow up for cardiac events.

A screening component to identify pre-clinical disease will include Holter ECG recordings and echocardiograms on patients without symptoms or evidence for heart disease seen in the SCI center during the course of the study and age-matched able-bodied veterans.

Hypothesis (a): The prevalence and incidence of cardiac diseases including coronary artery disease and cardiomyopathy will be higher in the SCI population than age-matched samples of the able-bodied population while valvular disease and arrhythmia will be similar. (b): The prevalence and incidence of cardiac disease in SCI individuals will be associated with level and completeness of injury (ie, higher occurrence in those with higher lesion levels and more complete injuries.) (c) The ECG will be helpful in SCI patients in early identification and secondary prevention of both ischemic and cardiomyopathic heart disease. (d) Continuous Holter ECG recordings or echocardiograms will only be indicated for screening specific SCI patients identified by clinical and electrocardiographic features.

ELIGIBILITY:
SCI patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800
Dates: Start 1999-10; Study Completion 2002-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Fryer, Ph.D. Asst. Director — Deprtment of Veterans Affairs, Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service; Nancy Rocheleau, Program Analyst — Department of Veterans Affairs, Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service
Locations (1):
- VAMC, Palo Alto, Palo Alto, California, United States